CLINICAL TRIAL: NCT03251495
Title: Immunologic Responses to a Live Attenuated Oral Cholera Vaccine
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Nadine Rouphael, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00097012; R01AI137127 (NIH)
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cholera
Keywords: Vaccination; Contagious Diseases; Tropical Medicine; Infectious Diseases
MeSH Terms: conditions — Cholera; Communicable Diseases | interventions — Vaxchora

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaxchora Vaccination (Experimental): Healthy participants will receive a single dose of oral live cholera vaccine.
  Interventions: Drug: Vaxchora

INTERVENTIONS:
Drug: Vaxchora — Vaxchora is a live attenuated cholera vaccine that provides immunity against V. cholerae serogroup O1. Participants will receive one single oral dose of 100 mL.

SUMMARY:
The primary objective of this study is to evaluate the antibody response to the cholera vaccine, Vaxchora®, in healthy subjects.

Investigators also seek to evaluate additional markers of the adaptive immune response including plasmablasts, activated B cells, memory B cells, and T cell responses in healthy subjects receiving cholera vaccine, produce monoclonal antibodies against cholera, and evaluate the safety and reactogenicity in healthy subjects receiving cholera vaccine.

DETAILED DESCRIPTION:
Vibrio cholerae causes an acute diarrheal disease responsible for more than 100,000 deaths and affects an estimated 3 to 5 million people annually. Recent epidemics in Haiti and Africa illustrate the continued reach of this pathogen. Across the globe, one billion people lack access to safe drinking water and are vulnerable to cholera. The increasing disease burden, and emergence of more virulent strains, suggest that more aggressive approaches to preventing cholera are needed. This includes renewed efforts to understand the mechanism of protective immunity against cholera and to improve the protective efficacy of current cholera vaccines.

Vaxchora is a live attenuated cholera vaccine that protects against some cholera strains. It has been approved by the FDA since June 2016. Since October, 2016, this vaccine has been recommended for certain travelers 18 through 64 years of age going to cholera-affected areas. The purpose of this study is to look at the immune responses to the FDA approved cholera vaccine (Vaxchora®).

This study aims to enroll 50 participants who will receive the Vaxchora live cholera vaccine, of whom 30 will undergo two procedures for small intestinal biopsies: one at screening and the other post vaccination (25 participants at Day 29 and 5 participants at day 90) by an upper endoscopy biopsy (EGD).

ELIGIBILITY:
Inclusion Criteria:

* Capable of informed consent and provision of written informed consent before any study procedures
* Capable of attending all study visits according to the study schedule
* Are in good health, as determined by medical history and targeted physical exam related to this history
* Female subjects of childbearing age must have a negative urine pregnancy test before study vaccination, and must use two forms of contraception to avoid pregnancy within one month of Vaxchora administration

Exclusion Criteria:

* Have an acute illness within 72 hours before vaccination
* Have any acute or chronic medical condition that, in the opinion of the principal investigator, would make vaccination unsafe or interfere with the evaluation of immune response to study vaccination
* Have a suppressed immune system as a result of illness, immunosuppressive medication, chemotherapy, or radiation therapy within 3 years prior to study vaccination
* Have taken oral or parenteral corticosteroids of any dose within 30 days before study vaccination
* Reside with individuals under the age of 2 or with an immunocompromised individuals
* Have a known history of autoimmune disease
* Have a history of Guillain-Barre Syndrome
* Have plans to receive any vaccine from 28 days prior to study vaccination until Day 29
* Has previously received a cholera vaccine or have a known history of V. Cholerae.
* Have donated blood or blood products within 56 days before study vaccination, plan to donate blood at any time during the 56-day duration of subject study participation, or plan to donate blood within 56 days after the last blood draw
* Have known hypersensitivity or allergy to any component of the vaccine or history of anaphylaxis with a vaccine or vaccine component
* Have allergy to tetracycline and/or ciprofloxacin
* Are pregnant or breastfeeding or plan to within one month of vaccination
* Traveled to a cholera endemic area and had traveler's diarrhea in the previous 5 years
* Have abnormal stool pattern (fewer than 3 stools/ week or greater than 2 stools/ day) or regular use of laxatives in the last 6 months
* Have current or recent antibiotic use in the past 14 days
* Are healthcare workers who have direct contact with patients who are immunocompromised, have unstable medical conditions, or are under the age of 2
* Are childcare caregivers who have direct contact with children who are 2 years or younger
* Are employed in the food industry
* Have received any vaccine within the previous 21 days
* History of bleeding disorders or current use of warfarin, aspirin, heparin, nonsteroidal anti-inflammatory drugs (NSAIDs) or other blood thinner/ anticoagulant medications in the past week for subjects undergoing intestinal biopsies.
* Use of benzodiazepines or narcotics for subjects undergoing intestinal biopsies 4 weeks prior to the procedure
* Any contraindications to endoscopy/concerns of the anesthesiologist for subjects who agree for esophagogastroduodenoscopy (EGD)/biopsies
* BMI > 35 kg/m^2
* Have a diagnosis of any small bowel disease. This includes but is not limited to inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, indeterminate colitis, or microscopic colitis), small bowel obstruction, celiac disease, h/o small bowel resection, small bowel lymphoma, Whipple's disease, primary Intestinal lymphangiectasis, abdominal radiation.
* Current medications for the treatment of Gastroesophageal reflux disease (GERD) or dyspepsia
* History of Helicobacter pylori (H. pylori) infection

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Level of Antibody Titers in Serum | Day 1 (pre-vaccination), Day 29
  Antibody response is evaluated as the level of antibody titers in serum.

SECONDARY OUTCOMES:
Plasmablast Levels | Days 1, 8, and 29
  Plasmablasts will be collected via blood draw and isolated and assessed for counts by the study team. A positive response is defined as a four-fold increase over the baseline measure.
Activated B Cell Levels | Days 1, 8, and 29
  Activated B cells will be collected via blood draw and isolated and assessed for counts by the study team. A positive response is defined as a four-fold increase over the baseline measure.
Memory B Cell Levels | Days 1 and 29
  Memory B cells will be collected via blood draw and isolated and assessed for counts by the study team. A positive response is defined as a four-fold increase over the baseline measure.
Correlation Between Antibody Titers and Plasmablasts, Activated B Cells, and Memory B Cells | Days 1 and 29
  The correlation between antibody titers and the level of plasmablasts, activated B cells, and memory B cells will be examined.
Number of Samples from which Monoclonal Antibodies Produced | Day 8
  The production of monoclonal antibodies against V. cholerae is assessed in a subset of participants.
Characterization of Monoclonal Antibodies Against V. Cholerae | Day 8
  The characterization of monoclonal antibodies against V. cholerae is assessed in a subset of participants.
Number of Adverse Events | Day 8, Day 29
  The number of solicited and unsolicited adverse events will be collected.
Number of Serious Adverse Events | Up to Day 365
  The number of serious adverse events will be collected during the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Rouphael, MD, Principal Investigator — Emory University
Locations (1):
- The Hope Clinic of Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adekunle O, Dretler A, Kauffman RC, Cho A, Rouphael N, Wrammert J. Longitudinal analysis of human humoral responses after vaccination with a live attenuated V. cholerae vaccine. PLoS Negl Trop Dis. 2021 Sep 3;15(9):e0009743. doi: 10.1371/journal.pntd.0009743. eCollection 2021 Sep. PMID 34478460

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT03251495/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT03251495/ICF_001.pdf